CLINICAL TRIAL: NCT04899284
Title: Impact of Early and Intensive Bimanual Stimulation on the Evolution of Bimanual Function in Infants With Clinical Findings Suggesting Unilateral Cerebral Palsy (BB-BIM)
Brief Title: Impact of Early Intensive Stimulation on Bimanual Function in Infants at High Risk of Unilateral CP (BB-BIM)
Acronym: BB-BIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Médico-Chirurgical de Réadaptation des Massues Croix Rouge Française (Other)
Collaborators: Groupement des Hôpitaux de l'Institut Catholique de Lille (GHICL) - France (Unknown); Hospices Civils de Lyon (Other); Laboratoire de Biomécanique et Mécanique des Chocs (LBMC) - France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB-BIM
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Cerebral Palsy
Keywords: Unilateral cerebral palsy; Unilateral brain lesion; Infantile cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infants eligible for Early Intensive Bimanual Stimulation (Experimental): Infants between 3 and 12 months of age at the time of inclusion, with unilateral brain injury and clinical signs of underuse of one of the two upper limbs
  Interventions: Other: Early Intensive Bimanual Stimulation

INTERVENTIONS:
Other: Early Intensive Bimanual Stimulation — Early intensive bimanual stimulation program for infants showing early signs of UCP, delivered by the family environment, in the child's familiar surroundings, under the guidance of a therapist, over a period of 2 months.

SUMMARY:
The aim of this study is to measure the impact of early bimanual stimulation in babies with clinical signs of underuse of one hand. The observation focuses on the developmental curve of hands use. The intervention is provided by the family environment and takes place in the child's familiar surroundings.

DETAILED DESCRIPTION:
Congenital hemiplegia, often referred to as Unilateral Cerebral Palsy (UCP), is characterized by a unilateral or asymmetrical brain injury that occurs around birth and impacts the development of manual skills and motor abilities of one side of the body.

Affected children frequently develop hemiplegia with major limitations in the use of their impaired hand, resulting in poor bimanual coordination, thus impacting the performance of daily activities at home, school and in the community.

Several intensive therapy approaches currently exist, including the bimanual approach (BIM) which aims to improve the use of the affected hand as an assisting hand in daily functional activities. These approaches have long been established as effective, however, with these children reaching 90% of their potential gross motor skills around the age of 5, or even earlier in some cases, there is a growing interest in earlier approaches, well before school age. It has also long been established that during the first year of life, there is a critical time frame for hand motor development.

The investigators have thus set up an intensive bimanual stimulation program for infants showing early signs of UCP, delivered by the family environment, in the child's familiar surroundings, under the guidance of a therapist, over a period of 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Baby between 3 and 12 months of age at the time of inclusion
* Clinical signs of underuse of one of the two upper limbs, (reported by the parents and authenticated by the HAI)
* Unilateral brain injury
* Brain imaging performed at birth or upon initial parental concerns
* Possibility of a home visit by the occupational therapist
* At least one parent volunteering to actively participate in the intensive stimulation
* Parental consent to enter the study
* Consent for image rights

Exclusion Criteria:

* Prematurity
* Lack of interest suggesting underlying associated disorders
* Active epilepsy

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Hand Assessment in Infants (HAI) | Change from baseline at 2 months with a weekly evaluation
  The HAI was developed for infants 3 to 12 months of age; the test is performed by filming the baby during a 10-minute play session. The examiner stimulates the baby with specific toys to induce hand actions, separately and together. Scoring includes 12 unimanual and five bimanual items, each scored on a 3-modality response scale (0, 1 or 2 points). The HAI provides a score for each of the upper limbs (out of 24 points), allowing quantification of possible asymmetry in the form of an index, as well as an interval measure of hand use (the total raw score out of 58 is converted to a scale from 0 to 100 points).

SECONDARY OUTCOMES:
Actimetry | Change from baseline at 2 months with a weekly evaluation
  The children will wear two accelerometers (one on each wrist) several times a week, during specific time sessions (training-game time guided by the parents and free play time). The data will be recorded on three axes (vertical, anteroposterior and mediolateral) and will be converted into activity quantity, with calculations such as the amplitude of the average vector, and the ratio of use between the two upper limbs.
Goal Attainment Scales | Change from baseline at 2 months with a weekly evaluation
  A maximum of 2 objectives will be determined with the parents: they will have to involve the use of the upper limb in practical situations of daily life, where a clear asymmetry of use has been observed, in order to be able to assess the evolution.
  The methodology used will be GAS 3 markers, the final score will be expressed on a 5-level ordinal scale, between (-2) and (+2), where (-2) corresponds to the initial level, (-1) to progress without having reached the expected level, (0) to reaching the expected level, (+1) to progress beyond the expected level, and (-2) to the most favourable result for the given objective.
Compliance | Change from baseline at 2 months with a weekly evaluation
  Interview reporting the number of bimanual stimulation sessions actually completed during the past week (from T6 to T13 during the intervention phase).
Parent satisfaction questionnaire | 2 months
  Assessment of satisfaction with the support provided by the occupational therapist, self-satisfaction with the role assigned to them, and satisfaction with the effectiveness of the program. List of questions to be answered with visual analog scales ranging from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Bard-Pondarré, OT, Principal Investigator — Croix rouge française Centre Médico-Chirurgical de Réadaptation des Massues. Lyon, France; Emmanuelle Chaléat-Valayer, PhD, Study Director — Croix rouge française Centre Médico-Chirurgical de Réadaptation des Massues. Lyon, France; Carole Vuillerot, PhD, Study Director — Hopital Femme Mère Enfant, l'Escale MPR pédiatrique (Hospices Civils de Lyon). Bron, France
Locations (1):
- Croix rouge française Centre Médico-Chirurgical de Réadaptation des Massues, Lyon, France

IPD SHARING:
Plan to Share IPD: No